CLINICAL TRIAL: NCT06854939
Title: Prospective Observational Study Using Personalized Minimal Residual Disease Assay (Signatera) to Evaluate the Kinetics and Detection Rate in Patients with Non-small Cell Lung Cancer
Brief Title: A Prospective Study Investigating the Relationship Between Minimal Residual Disease Detection, Monitoring Frequency, and Prognosis in Non-small Cell Lung Cancer Patients Eligible for Curative Treatment.
Acronym: MRDSEEKER
Status: Not yet recruiting | Type: Observational
Sponsor: National Cancer Center, Japan (Other Government)
Collaborators: Natera, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: JCOG2111A
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: NSCLC, Stage I, II, III
Keywords: Signatera™; minimal residual disease; MRD; lung cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm, Residual; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples With DNA — Blood samples collected in Streck tubes and EDTA tubes Tissue samples prepared on FFPE slides
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (4):
- Neoadjuvant therapy group: Resectable preoperative clinical stage II-III disease (with planned neoadjuvant therapy)
- Adjuvant therapy group: Resectable preoperative clinical stage IB-III disease (with no planned neoadjuvant therapy)
- Surgery-alone group: Resectable preoperative clinical stage IB-III disease (with no planned neoadjuvant therapy)
- Chemoradiotherapy group: Unresectable clinical stage III disease

SUMMARY:
Adding immune checkpoint inhibitors or molecularly targeted drugs as adjuvant therapy to curative treatments-such as surgery or chemoradiotherapy-for stage I-III non-small cell lung cancer (NSCLC) has been established as a standard of care and has improved treatment outcomes. However, there is currently no adequate method to determine which patients should receive these adjuvant therapies. Identifying those with a good prognosis without adjuvant therapy could reduce the risk of adverse events, lessen the burden of clinic visits, and reduce healthcare costs.

Among various approaches, ctDNA-based MRD (minimal residual disease) analysis is highly anticipated and has already been introduced into clinical practice for hematologic malignancies. However, solid tumors' development as a companion diagnostic has been limited, and regulatory approval is mainly being considered based on performance evaluation data. In this study, we will conduct a performance evaluation of MRD analysis using Signatera™ in patients with stage I-III NSCLC while also collecting other prognostic factors based on clinicopathological information and survival data.

ELIGIBILITY:
Inclusion Criteria:

1. A histopathologically confirmed diagnosis of non-small cell lung cancer (NSCLC)

   The diagnosis (by cytology or biopsy) must be one of the following: "adenocarcinoma," "squamous cell carcinoma," "non-small cell carcinoma consistent with adenocarcinoma," "non-small cell carcinoma consistent with squamous cell carcinoma," or "non-small cell carcinoma not otherwise specified (NOS)." If the histological subtype differs between cytology and biopsy specimens, the subtype determined by the biopsy specimen shall be used.

   At the time of enrollment, diagnoses of "squamous cell carcinoma" or "non-small cell carcinoma consistent with squamous cell carcinoma" are classified as squamous cell carcinoma, whereas "adenocarcinoma," "non-small cell carcinoma consistent with adenocarcinoma," and "non-small cell carcinoma NOS" are classified as non-squamous cell carcinoma.
2. Meets one of the following criteria (1-3):

1. Stage IB-III (preoperative clinical stage) deemed resectable, with no planned neoadjuvant therapy.

2. Stage III disease deemed amenable to curative-intent chemoradiotherapy. 3. Stage II-III (preoperative clinical stage) deemed resectable, with planned neoadjuvant therapy.

3) Age ≥ 18 years at the time of enrollment. 4) The attending physician has determined that tissue and blood samples can be provided.

5) Written informed consent has been obtained from the patient.

Exclusion Criteria:

* Presence of active multiple primary malignancies (defined as synchronous multiple cancers/tumors or metachronous multiple cancers/tumors with a disease-free interval of 3 years or less). However, even if the disease-free interval is less than 3 years, a history of clinical stage I prostate cancer or a completely resected cancer with any of the pathological stages specified below is not considered "active multiple primary malignancies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: non-small cell lung cancer (NSCLC)
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
2-year PFS | Analyses are planned to be performed 4.5 years after the start of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center Hospital, Chuo-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Undecided